CLINICAL TRIAL: NCT03826784
Title: A Multicenter, Randomized, Controlled, Blinded Study of the Efficacy and Safety of Bone Healing Accelerant Versus Standard of Care in Subjects With Open Tibia Fractures
Brief Title: Bone Healing Accelerant Versus Standard of Care for Open Tibia Fractures
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Combined into an international study (CAR-BHA-I21)
Sponsor: Carmell Therapeutics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAR-BHA-U31
Record Dates: First submitted 2019-01-29; First posted 2019-02-01 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2019-07

CONDITIONS: Tibial Fractures
MeSH Terms: conditions — Tibial Fractures | interventions — Butylated Hydroxyanisole

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- BHA (Experimental): Subjects treated with BHA + standard of care
  Interventions: Combination Product: BHA
- Control (No Intervention): Subjects treated as per standard of care

INTERVENTIONS:
Combination Product: BHA — BHA active ingredients include a blood-derived component and beta-tricalcium phosphate. It is applied directly to the bone fracture and nearby viable bone at the time of wound closure.
  Arms: BHA

SUMMARY:
This clinical study is being conducted to demonstrate the safety and effectiveness of the Bone Healing Accelerant (BHA) product when applied to tibia (leg bone) fractures with an external wound or skin break (also called open tibia fractures). It is hypothesized that by 6 months, the number of subjects with successful bone healing will be greater in the BHA-treated group compared to subjects treated with standard of care alone. Open tibia fractures were chosen for this study because healing rates are typically longer than for other bone fractures due to the limited vascular supply, limited soft tissue coverage, and higher risk of infection.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, subjects must meet all of the following criteria:

1. Patient is between the ages of 18-75 inclusive at time of randomization.
2. Patient has an acute open Gustilo-Anderson Type IIIA or IIIB fracture of the tibia shaft, with or without a fibula fracture, secondary to trauma.
3. Patient received antibiotic treatment within 2 hours of presentation at initial medical facility.
4. Patient underwent their first operative debridement within 24 hours of presentation at initial medical facility.
5. Patient is scheduled to have DWC within 14 days of initial injury.
6. The tibia fracture requires open fracture reduction and internal fixation with intramedullary (IM) nailing;

   * IM nailing has been cross-locked for stability with a 4-5mm interlock, with a minimum of 1 static screw above the fracture site and 1 static screw below the fracture site, and
   * All IM nails have a diameter between 8.5-12mm with 1.0-1.5mm over-reaming of the canal.

   The temporary use of external fixation prior to IM rodding and DWC is allowed.
7. Upon stabilization of the tibia fracture, the patient has a cortical deficit of less than or equal to 1.0cm involving no more than 50% of the tibia circumference. The cortical deficit of the residual 50% circumference must be less than 1.0cm. Gap assessments to be made with calibrated radiographs or visual inspection. In addition, patients are not likely to require a secondary procedure(s) to promote bone healing.
8. BHA is able to be applied through existing soft tissue defects created by the injury or those created during surgical treatment. No new incisions should be required specifically for application of BHA.
9. Patient is willing and able to comply with all study procedures including all pre-operative, post-operative and rehabilitation requirements.
10. Patient is able to give voluntary IC to participate and has signed an IC form specific to this study prior to study treatment and DWC.
11. Patients of childbearing potential must use adequate methods of contraception during the duration of follow-up (12-months). Adequate methods include abstinence, female and male sterilization, hormonal contraceptives, intrauterine devices (IUDs), implants, injectables, and double barrier methods.

Exclusion Criteria:

1. Patients who are currently participating in another investigational trial or having participated in a clinical investigation within the last 90 days or intend to during the course of the study.
2. Patients who are currently prisoners.
3. Patients who are unable to give informed consent.
4. Patients who are skeletally immature (<18 years of age or radiographic evidence of open tibial physes).
5. Patients with Type I, II, or IIIC open tibia fractures according to the Gustilo-Anderson classification.
6. Current injury is a pathological fracture.
7. Patients with additional injuries that could impact their ability to complete the required assessments and postoperative rehabilitation. Examples include but are not limited to the following:

   1. Head injury with impaired cognitive function,
   2. Spinal injury with resultant neurologic weakness or paralysis,
   3. Multi-trauma requiring prolonged hospitalization or recovery that, in the opinion of the investigator, the treatment and/or rehabilitation of such injuries will substantially interfere with the treatment, rehabilitation or other requirements outlined in this protocol,
   4. Concomitant ipsilateral or contralateral lower extremity injury/fracture(s) if, in the opinion of the investigator, the treatment and/or rehabilitation of such fracture(s) will substantially interfere with the treatment, rehabilitation or other requirements outlined in this protocol.
   5. Sustained severe burns (>10% total body surface area [TBSA] or >5% TBSA with full thickness or circumferential injury)
   6. Compartment syndrome of the leg diagnosed preoperatively
8. Patients with pre-existing conditions, mental/psychosocial disorders, or who are taking medication that may delay or impair the fracture healing process or that could impact their ability to return for follow-up visits and/or complete the required assessments and postoperative rehabilitation. Examples include but are not limited to the following:

   1. Renal insufficiency with serum creatinine of 3.5 mg/dL or higher or being treated with renal dialysis,
   2. Uncontrolled diabetes mellitus with A1C of greater than or equal to 10%,
   3. Serum Aspartate Aminotransferase (AST) greater than 2 times the upper limit of normal or diagnosed hepatitis C or hepatitis B,
   4. Neurological or neuromuscular disorders affecting ambulatory capability or cognition, such as Parkinson's disease, myasthenia gravis, or stroke with relevant residual neurological deficit,
   5. Current medications that could interfere with fracture healing such as systemic corticosteroids,
   6. Morbid Obesity with BMI greater than or equal to 40 kg/m2,
   7. A current endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's disease, renal osteodystrophy, hyperthyroidism, parathyroid hormone disorder, Ehler-Danlos syndrome, osteogenesis imperfecta, or Cushing's disease),
   8. History of osteomyelitis of index lower extremity or evidence of active soft tissue or bone infection at this site of injury at the time of DWC,
   9. Patients with immune deficiency or history of auto-immune disease.
9. Patients with an active malignancy or a history of any invasive malignancy (except non-melanoma skin cancer), unless the patient has been treated with curative intent and there have been no clinical signs or symptoms of malignancy for at least 5 years.
10. Patients with any medical condition or life circumstances that in the surgeon's opinion could impact their ability to return for follow-up visits and/or complete the required assessments and postoperative rehabilitation. Examples include but are not limited to the following:

    1. Patient lives too far away making the return for study visits to the surgeon's facility unlikely,
    2. The patient has known alcohol or drug abuse within 3 months of screening to a degree that makes it unlikely the patient will follow study requirements.
11. Patients who are known to have anaphylactic or severe systemic reaction to human blood products, genipin, β-TCP, glycerin or to other components of the investigative product formulation.
12. Female patients of child-bearing potential who meet any of the following criteria:

    * Patient is currently pregnant (prior diagnosis or a positive pregnancy test at baseline), or planning to become pregnant any time during the course of the study
    * Currently breastfeeding or planning to breastfeed at any time during the course of the study
13. Upon stabilization of the tibia fracture, the patient has a bone gap greater than 1.0cm apparent by calibrated radiographs or by visual inspection and/or the patient is highly likely to require secondary intervention procedure(s), surgical or nonsurgical (e.g., bone stimulation or ultrasound treatment) for the index fracture.
14. Patients who have mal-alignment post-IM nailing of >10° in the coronal plane or >15° in the sagittal plane.
15. Patients who received only plates and screws for tibia fracture stabilization.
16. At the time of the DWC surgery, patients who have a planned secondary intervention procedure, surgical or nonsurgical (e.g., bone stimulation or ultrasound treatment) for the index fracture.
17. Patients being treated with any form of local antibiotics at the time of DWC.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Composite healing measure | 6 months
  Proportion of subjects in each arm meeting the healing success criteria. A binary (Yes/No) outcome for overall healing will be derived from the following three outcomes: Radiographic healing as measured by a score of at least 13 on the modified Radiographic Union Scale in Tibia fractures (mRUST, range bad to good 1-16), ambulation as measured by a score of at least 2 on the Function IndeX for Trauma scale (range bad to good 0-3), and no secondary intervention to promote bone healing. All three components must be met for a "yes" on composite healing.

SECONDARY OUTCOMES:
Radiographic healing | 6 months
  Population mean Modified Radiographic Union Scale in Tibia Fractures (mRUST) scores (range bad to good is 4-16)
Secondary intervention (surgical or nonsurgical) | 6 months
  Proportion of subjects not having secondary intervention conducted specifically to promote bone healing needed
Surgical site infection | 12 months
  Proportion of subjects having surgical site infection through 12 months as determined by CDC guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Janet M Vargo, PhD, Study Director — Carmell Therapeutics
Locations (1):
- Carmell Therapeutics, Pittsburgh, Pennsylvania, United States